CLINICAL TRIAL: NCT00890357
Title: Identifying Factors Underlying the Discontinuation of Triptans
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Todd J. Schwedt, PI, Mayo Clinic
Other Study IDs: 09-0111
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Migraine; Medication Adherence
MeSH Terms: conditions — Migraine Disorders; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Triptan User
- Triptan Discontinued

SUMMARY:
The objective of this study is to identify reasons migraine patients stop using triptan medications for abortive headache treatment. It is hypothesized that inadequate education of the patient at the time of prescribing the triptan is positively associated with triptan discontinuation.

ELIGIBILITY:
Triptan User Inclusion Criteria:

* Episodic Migraine or Chronic Migraine
* Have used a triptan medication in the prior 3 months
* Have used triptan medications for at least 1 year

Triptan Discontinuation Inclusion Criteria:

* Episodic Migraine or Chronic Migraine
* Used any triptan medication in the last 2 years
* Have not used a triptan medication in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Specialty Headache Clinics
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schwedt, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of South Florida College of Medicine, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Derived] Wells RE, Markowitz SY, Baron EP, Hentz JG, Kalidas K, Mathew PG, Halker R, Dodick DW, Schwedt TJ. Identifying the factors underlying discontinuation of triptans. Headache. 2014 Feb;54(2):278-89. doi: 10.1111/head.12198. Epub 2013 Sep 3. PMID 24001117